CLINICAL TRIAL: NCT00941161
Title: Effect of Oral Combination Therapy of Metformin Extended Release Over Glimepiride in a Single Dosage Form in Patients With Type 2 Diabetes Mellitus With Failure of Monotherapy
Brief Title: Effect of Oral Combination Therapy in a Single Dosage Form in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Jorge Gonzalez Canudas, M.D., Laboratorios Silanes, S.A. de C.V.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DMGlime-04
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; glimepiride

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- combination (Experimental): long acting Metformin/Glimepiride
  Interventions: Drug: metformin/glimepiride combination
- metformin (Active Comparator): metformin hydrocloride
  Interventions: Drug: metformin
- glimepiride (Active Comparator): glimepiride
  Interventions: Drug: glimepiride

INTERVENTIONS:
Drug: metformin/glimepiride combination — long acting metformin/glimepiride 1g/2mg
  Arms: combination
Drug: metformin — long acting metformin 1g once a day with fasting glucose 130-199mg/dL or long actin metformin 1g twice a day (before dinner and before breakfast) with fasting glucose 200-270mg/dL
  Arms: metformin
Drug: glimepiride — glimepiride 2mg once a day with fasting glucose 130-199mg/dL, or glimepiride 2mg twice a day (before dinner and before breakfast) with fasting glucose 200-270mg/dL
  Arms: glimepiride

SUMMARY:
The aim of the study is to determinate the effect of combined oral therapy of long acting metformin/glimepiride in a single dose in patients with type 2 diabetes mellitus and monotherapy failure.

DETAILED DESCRIPTION:
A randomized double-blind clinical trial, to determine the effect of combined therapy of oral prolonged-release metformin/glimepiride in a single dosage form on fasting glucose and HbA1c. Patients will be included in this study are patients with diabetes mellitus and secondary failure to monotherapy. Will also assess the effect of combined therapy on the oral lipid profile (total cholesterol, LDL, HDL, VLDL, Triglycerides) and on the sensitivity and insulin secretion. We evaluate the clinical measurements, laboratory and safety during 3 months, through the allocation of subjects to three study groups (metformin, glimepiride and metformin extended release / glimepiride)

ELIGIBILITY:
Inclusion Criteria:

* 40 to 65 years old
* Ability to communicate and to meet the requirements of the study
* Signed Written Informed Consent before to conducting any study
* Body Mass Index (BMI) = 25-40kg/m2
* Stable weight in the past three months (variability <5%)
* Meal plan and monotherapy with oral hypoglycaemic fails
* Fasting glucose = 130-270 mg/dL
* HbA1c > 7%
* isocaloric diet with a minimum of 250 grams of carbohydrates per day in the three days prior to making the laboratory tests

Exclusion Criteria:

* Suspected or confirmed pregnancy
* Nursing
* Inability to secure the non-pregnant during the study duration
* Hypersensitivity to any of the drugs under study
* Treatment with oral hypoglycemic or insulin
* Consumption of substance with toxic effects on any organ system
* Liver failure, heart failure, kidney failure or thyroid disease
* Chronic intake of alcohol
* Periods of acute or chronic diarrhea or vomiting
* Consumption of antifungal azoles, MAO inhibitors, nifedipine,furosemide, amiloride, digoxin, procainamide, quinidine, quinine, triamterene and vancomycin

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
fasting glucose, HbA1c | three months

SECONDARY OUTCOMES:
total cholesterol, C-LDL, C-HDL, triglycerides, VLDL, insulin | three months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Gonzalez, M.D., Master, Study Director — Laboratorios Silanes S.A. de C.V.; Manuel Gonzalez, Ph.D., Study Chair — University of Guadalajara; Esperanza Martínez, Ph.D., Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Ciencias de la Salud. Universidad de Guadalajara, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] International Diabetes Federation / International Association for the Study of Obesity. Diabetes and Obesity 11-21, 2004
- [Background] Grundy SM, Pasternak R, Greenland P, Smith S Jr, Fuster V. AHA/ACC scientific statement: Assessment of cardiovascular risk by use of multiple-risk-factor assessment equations: a statement for healthcare professionals from the American Heart Association and the American College of Cardiology. J Am Coll Cardiol. 1999 Oct;34(4):1348-59. doi: 10.1016/s0735-1097(99)00387-3. No abstract available. PMID 10520820
- [Background] Tseng KH. Standards of medical care in diabetes--2006: response to the American Diabetes Association. Diabetes Care. 2006 Nov;29(11):2563-4; author reply 2564-5. doi: 10.2337/dc06-0805. No abstract available. PMID 17065711
- [Background] Cohen J, Colman P. Type 2 diabetes--the pharmacotherapy of glycaemic control and risk factor modification. Aust Fam Physician. 2006 Jun;35(6):380-4. PMID 16751851
- [Background] Nathan DM, Buse JB, Davidson MB, Heine RJ, Holman RR, Sherwin R, Zinman B; Professional Practice Committee, American Diabetes Association; European Association for the Study of Diabetes. Management of hyperglycaemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy. A consensus statement from the American Diabetes Association and the European Association for the Study of Diabetes. Diabetologia. 2006 Aug;49(8):1711-21. doi: 10.1007/s00125-006-0316-2. No abstract available. PMID 16802130
- [Background] Riddle M. Combining sulfonylureas and other oral agents. Am J Med. 2000 Apr 17;108 Suppl 6a:15S-22S. doi: 10.1016/s0002-9343(00)00338-7. PMID 10764846
- [Background] Bermudez-Pirela VJ, Cano C, Medina MT, Souki A, Lemus MA, Leal EM, Seyfi HA, Cano R, Ciscek A, Bermudez-Arias F, Contreras F, Israili ZH, Hernandez-Hernandez R, Valasco M. Metformin plus low-dose glimeperide significantly improves Homeostasis Model Assessment for insulin resistance (HOMA(IR)) and beta-cell function (HOMA(beta-cell)) without hyperinsulinemia in patients with type 2 diabetes mellitus. Am J Ther. 2007 Mar-Apr;14(2):194-202. doi: 10.1097/01.pap.0000249909.54047.0e. PMID 17414590
- [Background] Gonzalez-Ortiz M, Martinez-Abundis E; Grupo para el Tratamiento de la Diabetes Mellitus con Combinaciones. [Efficacy and safety of glimepiride plus metformin in a single presentation, as combined therapy, in patients with type 2 diabetes mellitus and secondary failure to glibenclamide, as monotherapy]. Rev Invest Clin. 2004 May-Jun;56(3):327-33. Spanish. PMID 15612515
- [Background] Mandal U, Gowda V, Ghosh A, Selvan S, Solomon S, Pal TK. Formulation and optimization of sustained release matrix tablet of metformin HCl 500 mg using response surface methodology. Yakugaku Zasshi. 2007 Aug;127(8):1281-90. doi: 10.1248/yakushi.127.1281. PMID 17666882
- [Background] Schwartz S, Fonseca V, Berner B, Cramer M, Chiang YK, Lewin A. Efficacy, tolerability, and safety of a novel once-daily extended-release metformin in patients with type 2 diabetes. Diabetes Care. 2006 Apr;29(4):759-64. doi: 10.2337/diacare.29.04.06.dc05-1967. PMID 16567811
- [Background] Bailey CJ, Turner RC. Metformin. N Engl J Med. 1996 Feb 29;334(9):574-9. doi: 10.1056/NEJM199602293340906. No abstract available. PMID 8569826
- [Background] McCall AL. Clinical review of glimepiride. Expert Opin Pharmacother. 2001 Apr;2(4):699-713. doi: 10.1517/14656566.2.4.699. PMID 11336617
- [Background] Schneider J. An overview of the safety and tolerance of glimepiride. Horm Metab Res. 1996 Sep;28(9):413-8. doi: 10.1055/s-2007-979829. PMID 8911975